CLINICAL TRIAL: NCT05588310
Title: Quantification of the Socio-economic Multifacet Burden of Alopecia Areata and Identification of the Associated Factors
Acronym: PelBurd
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0054; 2022-A00986-37 (Other: ID-RCB Number)
Record Dates: First submitted 2022-06-10; First posted 2022-10-20 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Alopecia Areata
Keywords: Socio-economic burden; alopecia areata; out-of-pocket expenditures
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Alopecia areata (AA) is a complex autoimmune disorder with an estimated lifetime risk of 1.7% where both genetic pre-disposition and environmental factors contribute. It typically presents with sharply demarcated round patches of non-scarring hair loss that may present at any age. Many patients with AA are dissatisfied with current medical treatments and use alternative therapies and cosmetics. This study will generate new data on the current situation of psychosocial and financial burden of AA. It will help to identify unmet needs and to understand the disease issues. It will also be the basis for the planification of future supporting measures.

DETAILED DESCRIPTION:
Alopecia areata (AA) is a complex autoimmune disorder with an estimated lifetime risk of 1.7% where both genetic pre-disposition and environmental factors contribute. It typically presents with sharply demarcated round patches of non-scarring hair loss that may present at any age. Current medical therapies (topical or systemic) for AA are not reliably effective, particularly for severe disease and there is no robust evidence from high-quality randomized controlled trials. Patients with AA experience significant mental health and health related quality of life (HRQoL) impairment. Furthermore, at the country level, skin conditions such as AA ranged from 2nd to 11th leading cause of years lived with disability. It was shown that AA appears to affect all countries across the world similarly, and the health burden has remained stable despite substantial advances in healthcare and health-related resources. More recently, Mesinkovska et al demonstrated that the impact of AA extends beyond cosmetic concerns and carries a considerable psychosocial burden.

Many patients with AA are dissatisfied with current medical treatments and use alternative therapies and cosmetics. Cosmetics and not reimbursed treatments can weigh heavily on patients spending.This study will generate new data on the current situation of psychosocial and financial burden of AA. It will help to identify unmet needs and to understand the disease issues. It will also be the basis for the planification of future supporting measures.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years).
* Alopecia Areata whose diagnosis has been confirmed by a dermatologist according to the standardized diagnostic criteria.
* < 2 years duration of current episode of scalp hair loss.
* Severity > S2 (> 25% hair loss) as assessed by the Alopecia Tool (SALT).

Exclusion Criteria:

* Patients under juridical protection.
* Patients not covered by social security.
* Patients unable to understand French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients whom suffer from Alopecia Areata
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Calculate the Out Of Pocket (OOP) expenditures of patients whom suffer from alopecia areata | 12 months
  To describe the OOP expenditures related to Alopecia Areata from a patient point of view by using the retrospective questionnaire during 6 months and using the prospective weekly follow-up patient diary during 6 months.

SECONDARY OUTCOMES:
Calculate direct medical costs and indirect costs limited to work stopping and working reduction time related to Alopecia Areata | 12 months
  To describe direct medical costs, hospitalizations stays, visits and additional tests will be collected using patients diary and interviews. These data will be completed by PMSI (Programme de Médicalisation des Systèmes d'Information) data of each participating hospital. Indirect costs will be limited to work stopping or working reduction time and will be collected by self reporting PelBurd Version n°2.0 of April 8, 2022 10 in patients diaries. Socio-professional category and job will be collected during the first visit in order to assess costs related job changes. These costs will be established over a period of one year on retrospective (interview) and prospective (diary) basis.
Evaluate the impact of Alopecia Areata on Health Related Quality of Life (HRQoL) - DLQI | 6 months
  Health Realted Quality of Life will be assessed using the validated French versions of the dermatology specific questionnaire " Dermatology Life Quality Index " (DLQI). The questionnaire will be self-evaluated by patients at M0 and M6. DLQI consists of 10 questions with 4 points likert answers and ranges from 0 (no effect on QoL) to 30 maximum effect on QoL. DLQI scores can also be categorised into 5 different levels (very much, a lot, a little, not at all, not relevant) 13.
Evaluate the impact of Alopecia Areata on Health Related Quality of Life (HRQoL) - AA-QLI | 6 months
  Health Realted Quality of Life will be assessed using the validated French versions of the disease specific questionnaire for AA (AA-QLI). The questionnaire will be self-evaluated by patients at M0 and M6. AA-QLI consists of 21 questions with 4 points likert answers. It is scored by averaging 3 subscales and presented on a 0 (no effect on QoL) to 100 points scale.
Evaluate the patient's perceived stress | 6 months
  Evaluate the patient's perceived stress by using the validated French version of the Perceived stress scale (PSS) self-evaluated by patients at M0 and M6. The perceived stress scale consisted of 10 questions with 5 points likert answers. It ranges from 0 (no perceived stress) to 40 (highest possible perceived stress) and can be categorized into 3 different levels (low, moderate and high perceived stress)
Evaluate the impact of Alopecia Areata on depression symptoms | 6 months
  Evaluate the impact of Alopecia Areata on depression symptoms by using the validated French version of the Patient health questionnaire 9 (PHQ-9). This questionnaire will be self-evaluated by patients at M0 and M6. The PHQ9 questionnaire consists of 9 questions with 4 points likert answers and ranges from 0 (absence of depressive symptoms) to 27 (severe depressive symptoms). PHQ-9 scores can be categorized in 5 levels (none, mild, moderate, moderately severe, severe). Patients with a PHQ-9 score above 10 should be referred to a psychiatric evaluation.
Evaluate the impact of Alopecia Areata on anxiety symptoms | 6 months
  To evaluate the impact of AA on anxiety symptoms by using the validated French version of the General anxiety disorder 7 (GAD 7), self-evaluated by patients at M0 and M6. The GAD-7 consists of 7 questions with 4 points likert answers and ranges from 0 (absence of anxious symptoms) to 27 (severe anxious symptoms). GAD-7 scores can be categorized in 4 levels (none, mild, moderate, severe).
Describing the care pathway for Alopecia Areata patients | 6 months
  To describe the care pathway for Alopecia Areata patients (delay to diagnosis and treatment), the clinician will report during the first consultation (M0), the number of consulted physicians and the following dates: first symptoms, first appointment with a medical doctor (MD), first appointment with a dermatologist, diagnosis, beginning of the first treatment. In rare or neglected diseases diagnostic delay is usually defined as the delay between first consultation with a MD and the final diagnosis . We will also calculate the delay to consultation (defined as the time between first symptoms and first consultation with a MD), the delay to dermatologist consultation (defined as the time between first consultation with a MD and first consultation with a dermatologist) and the delay to first treatment (defined as the time between the first consultation with a MD and the first treatment).
Describing the impact of Alopecia Areata on work productivity | 6 months
  To describe the impact of AA on work productivity, we will use the validated French version of the Work Productivity and Activity Impairment (WPAI) (self-assessed by patients at M0 and M6). The WPAI is a 6 questions score that assesses hours missed at work, loss of productivity at work and in daily activities because of a specific health issue. The WPAI is expressed as 4 impairments: percent work time missed due to health, percent impairment while working due to health issue, percent overall work impairment due to health issue, percent activity impairment due to health issue

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Mazereeuw-Hautier, Pr, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse University hospital, Toulouse, France